CLINICAL TRIAL: NCT04969224
Title: A Phase 3b Open-label Study Evaluating the Effects of Elexacaftor/Tezacaftor/Ivacaftor on Cough and Physical Activity in Cystic Fibrosis Subjects 12 Years of Age and Older Who Are Heterozygous for the F508del Mutation and a Minimal Function Mutation (F/MF)
Brief Title: A Study to Evaluate ELX/TEZ/IVA on Cough and Physical Activity in Participants With Cystic Fibrosis (CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX20-445-126; 2021-001628-16 (EudraCT Number)
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Results first posted 2023-10-03 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ELX/TEZ/IVA (Experimental): Participants received ELX 200 milligram (mg) once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the treatment period approximately 13 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed dose combination (FDC) tablet for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the effects of elexacaftor/tezacaftor/ivacaftor (ELX/TEZ/IVA) on cough and physical activity using wearable technology in CF participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Forced expiratory volume in 1 second (FEV1) value ≥30% and ≤90% predicted
* Heterozygous for CF transmembrane conductance regulator gene (CFTR) F508del mutation and a minimal function mutation (F/MF genotypes)

Key Exclusion Criteria:

* Clinically significant liver cirrhosis
* Solid organ or hematological transplantation
* Non-ambulatory status
* Lung infection with organisms associated with a more rapid decline in pulmonary status

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (19):
- Australia (8):
  - Royal Adelaide Hospital, Adelaide
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne, VIC
  - Institute for Respiratory Health, Nedlands
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville, VIC
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
- Belgium (4):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (3):
  - University of Calgary Medical Clinic of the Foothills Medical Centre, Calgary
  - University of Alberta Hospital, Edmonton Clinic, Edmonton
  - Queen Elizabeth II Health Sciences Center, Halifax
- Spain (4):
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Corporacio Sanitaria Parc Tauli - Sabadell Hospital Universitari, Sabadell

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was conducted in participants with cystic fibrosis, aged 12 years and older, who are heterozygous for the F508del mutation and the minimal function mutation (F/MF) genotypes.
Groups:
- ELX/TEZ/IVA: Participants received elexacaftor (ELX) 200 milligram (mg) once daily (qd)/ tezacaftor (TEZ) 100 mg qd/ ivacator (IVA) 150 mg every 12 hours (q12h) in the treatment period approximately 13 weeks.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA
Started | 82
Completed | 80
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Enrolled but never dosed | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug during the treatment period were included in the baseline analysis.
Groups:
- ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period approximately 13 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 78
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 81
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction From Baseline in Cough Frequency (Cough Events Per Day) to the Average of Week 8 Through Week 12
Description: Percent reduction in cough frequency was analyzed with a mixed effects model for repeated measures (MMRM), with change from baseline at each post-baseline visit on the natural log scale as the dependent variable. The percent reduction was estimated as 100% × (1-exponential form of LS mean change estimate from the MMRM).
Time Frame: Baseline, Week 8 through Week 12
Population: The Full Analysis Set (FAS) will include all enrolled participants who carry the intended CFTR allele mutation and have received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent reduction
Groups:
- ELX/TEZ/IVA: Participants received ELX 200 mg qd/ TEZ 100 mg qd/ IVA150 mg q12h in the treatment period approximately 13 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 80
percent reduction | 91.7 [89.2 to 93.6]

2. Secondary Outcome: Absolute Change From Baseline in Total Step Count Per Day to the Average of Week 8 Through Week 12
Time Frame: Baseline, Week 8 through Week 12
Population: FAS. Here, "Overall Number of Participants Analyzed" signifies participants who were evaluable for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: step count per day
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 80
step count per day | 637.56 [298.16 to 976.96]

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 17
Description: Safety Set included all participants who had received at least 1 dose of study drug.
Arm/Group | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/81
Serious Adverse Events (participants affected / at risk) | 2/81
Other Adverse Events (participants affected / at risk) | 56/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=81)
Pancreatitis (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=81)
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 11
COVID-19 (Infections and infestations) | 13
Nasopharyngitis (Infections and infestations) | 13
Upper respiratory tract infection (Infections and infestations) | 7
Headache (Nervous system disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT04969224/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/24/NCT04969224/SAP_001.pdf